CLINICAL TRIAL: NCT01520935
Title: Burden of Influenza in the United Kingdom, 1996-2008
Brief Title: Influenza Burden Assessment in the United Kingdom, 1996-2008
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Sage Analytica (Industry)
Responsible Party: Sponsor
Other Study IDs: 116273
Record Dates: First submitted 2012-01-23; First posted 2012-01-30 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Influenza
Keywords: Office of National Statistics; Burden of Disease; Influenza; Hospital Episode Statistics; General Practitioners Research Database
MeSH Terms: conditions — Influenza, Human | interventions — Data Collection

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Cohort Group
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The study, will use four primary data sources: the General Practice Research Database (GPRD, for mild outcomes), the Hospital Episode Statistics database (HES, for hospitalizations), the Office of National Statistics mortality database (ONS, for mortality), and weekly virology data from the Health Protection Agency (HPA).
  Weekly time series of the rates of various influenza-related health outcomes in the various databases, such as office visits for acute otitis media and hospitalizations for pneumonia will be constructed. Statistical models, guided by weekly numbers of cases of laboratory-confirmed influenza and respiratory syncytial virus (RSV) contained in the HPA virology data, to estimate the portions of the various outcomes that can be attributed to influenza will be constructed. Finally, the seasonal impact of influenza by risk status, vaccination status, and seasons in which a well-matched versus mismatched influenza vaccine was used, will be assessed.

SUMMARY:
The study will assess the burden of influenza by age, risk status, vaccination status and influenza subtype, in order to create a complete profile of the burden of influenza-related morbidity and mortality in United Kingdom from 1996 to 2008.

DETAILED DESCRIPTION:
This epidemiological study is a modelling of time series retrospectively extracted from multiple databases. The data collection will be a query of existing electronic healthcare databases.

ELIGIBILITY:
Inclusion Criteria:

• Registration with an acceptable flag in the GPRD, or registration with a potentially influenza-related event in the HES database or the ONS mortality data.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People of any age in the United Kingdom who were registered with an acceptable flag in the GPRD, or with a potentially influenza-related event in the HES database or the ONS mortality data.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Incidence of medically attended health outcomes (~20 relevant mild and severe) related to influenza | From 1996 to 2008 (up to 13 years)
Relative impact of influenza on high versus low risk populations | From 1996 to 2008 (up yo 13 years)
Relative impact of influenza during match versus mismatched seasons | From 1996 to 2008 (up to 13 years)
Relative impact of influenza on vaccinated versus unvaccinated populations | From 1996 to 2008 (up to 13 years)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Matias G, Taylor RJ, Haguinet F, Schuck-Paim C, Lustig RL, Fleming DM. Modelling estimates of age-specific influenza-related hospitalisation and mortality in the United Kingdom. BMC Public Health. 2016 Jun 8;16:481. doi: 10.1186/s12889-016-3128-4. PMID 27278794
- [Derived] Fleming DM, Taylor RJ, Haguinet F, Schuck-Paim C, Logie J, Webb DJ, Lustig RL, Matias G. Influenza-attributable burden in United Kingdom primary care. Epidemiol Infect. 2016 Feb;144(3):537-47. doi: 10.1017/S0950268815001119. Epub 2015 Jul 13. PMID 26168005